CLINICAL TRIAL: NCT04035551
Title: Health Evaluation And Learning for Total Parenteral Nutrition (TPN) at Home (HEALTH)
Brief Title: Health Evaluation And Learning for Total Parenteral Nutrition (TPN) at Home Patient Registry
Acronym: HEALTH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coram Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CT-10-06
Record Dates: First submitted 2019-07-09; First posted 2019-07-29 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-03

CONDITIONS: Malnutrition; Patients Requiring Home Parenteral Nutrition
Keywords: Home; HPN; Homecare
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients receiving home parenteral nutrition: Includes patients receiving home parenteral nutrition for any indication.

SUMMARY:
The HEALTH Registry is a prospective, observational, non-interventional registry study of patients receiving home parenteral nutrition therapy in the US for a variety of indications.

DETAILED DESCRIPTION:
The objective of the HEALTH Patient Registry is to establish and track therapy utilization and outcomes of patients receiving home parenteral nutrition therapy. Data collected will include information on patient safety, clinical outcomes, resource utilization and health-related quality of life (QOL). The goals of this Registry include:

* To better understand the patients and populations requiring HPN in the U.S.
* To measure clinical outcomes associated with HPN
* To identify areas for focused quality improvement interventions
* To provide opportunity for resource allocation identification and improvement

ELIGIBILITY:
Inclusion Criteria:

* Patient of any age, gender, and indication referred to Coram/CVS Specialty Infusion Services to receive HPN in an alternate site of care, such as the home or infusion suite
* Patient must be managed by Coram/CVS Specialty Infusion Services
* The patient or the patient's caregiver must be willing to receive care and comply with the teaching and training necessary to administer treatment

Exclusion Criteria:

* Patient is unable to start, or stops receiving HPN
* Patient is NOT managed by Coram/CVS Specialty Infusion Services
* A patient and/or a patient's insurance will not cover cost of HPN therapy with Coram/CVS, or a patient elects not to start treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The HEALTH Registry program will collect data representative of patients receiving total parenteral nutrition (TPN) in the homecare setting.
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life over time: The Short Form (36) | At baseline and every 6 months during therapy through study completion, up to 3 years
  To examine the effect of HPN support on quality of life (functional health and well-being) as measured by The Short Form (36) Health Survey (SF-36v2). Physical component summary (PCS) and mental component summary (MCS) scores on a scale of 0 to 100 with higher scores reflecting better outcomes will be utilized.
Efficacy of Home Parenteral Nutrition defined as the percentage of patients reaching their PN therapy goals | through study completion, an average of 3 years
  The therapy goals (i.e. weight gain, weight loss, weight maintenance, resolution of GI issue, etc). will be recorded at study start. Percentage of patients reaching their designated therapy goal will be recorded (presented as a single percentage of patients that successful reached any therapy goal)

SECONDARY OUTCOMES:
Catheter-related infections | through study completion, an average of 3 years
  Determine rate of catheter-related blood stream infections (CRBSIs) ( per 1000 catheter days)
Number of hospital readmissions and ER visits | through study completion, an average of 3 years
  Assess number of hospital readmissions and visits to the ER
Mortality rate | through study completion, an average of 3 years
  Number of study participants who expired during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeLegge, MD, Principal Investigator — Coram
Locations (1):
- Coram CVS Specialty Infusion Services, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: No